CLINICAL TRIAL: NCT00054808
Title: A Phase II Multicenter Study of Gallium Nitrate in Patients With Relapsed or Refractory Non-Hodgkin's Lymphoma
Brief Title: Phase II Gallium Nitrate in Relapsed or Refractory Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genta Incorporated (Industry)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: Genta-GGN202
Record Dates: First submitted 2003-02-10; First posted 2003-02-13 (Estimated); Last update posted 2006-02-08 (Estimated); Status verified 2006-02

CONDITIONS: Non-Hodgkin's Lymphoma; Relapsed Lymphoma; Refractory Lymphoma; Low-Grade Lymphoma; Intermediate-Grade Lymphoma
Keywords: Gallium Nitrate; Ganite; NHL; Relapsed
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma; Recurrence | interventions — gallium nitrate

INTERVENTIONS:
Drug: gallium nitrate

SUMMARY:
Eligible patients will have low- or intermediate-grade Non-Hodgkin's Lymphoma (NHL) that has progressed after standard chemotherapy. Patients will receive gallium nitrate 300 mg/m2/day by continuous IV infusion for 7 consecutive days using a portable infusion pump. Hospitalization is not required. Stable or responding patients will receive additional gallium nitrate infusions every 3 weeks until the time of disease progression, for a maximum total of 8 infusions, or 2 cycles after complete remission has been documented.

DETAILED DESCRIPTION:
This study seeks to define the role of gallium nitrate in a specific population of patients who are expected to have received prior therapy. Preliminary clinical studies have suggested substantial evidence of antitumor activity in patients with relapsed or refractory non-Hodgkin's Lymphoma treated with gallium nitrate.

ELIGIBILITY:
Low- or intermediate-grade NHL using the International Working Formulation, subtypes IWF A-G:

Using the Updated REAL/WHO Classification, the following pathologic subtypes are eligible:

* Small lymphocytic lymphoma
* Lymphoplasmacytic lymphoma/immunocytoma
* Follicular lymphoma
* Diffuse large B-cell lymphoma
* Peripheral T-cell lymphoma, not otherwise characterized

Progression of disease following treatment with standard chemotherapy

Bi-dimensionally measurable disease

Performance Status: ECOG < = 2

Patients with mantle cell lymphoma or mycosis fungoides are not eligible

Patients with known history of CNS metastasis are not eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2002-06

CONTACTS AND LOCATIONS:
Locations (1):
- Genta, Berkeley Heights, New Jersey, United States

REFERENCES:
- [Background] Warrell RP Jr, Coonley CJ, Straus DJ, Young CW. Treatment of patients with advanced malignant lymphoma using gallium nitrate administered as a seven-day continuous infusion. Cancer. 1983 Jun 1;51(11):1982-7. doi: 10.1002/1097-0142(19830601)51:113.0.co;2-l. PMID 6839291